CLINICAL TRIAL: NCT06337175
Title: Predictors of Post-alteplase Different Subtypes of Hemorrhagic Transformation of Brain Infarction in the Middle East
Brief Title: Predictors of Post-alteplase Hemorrhagic Transformation of Brain Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, principal investigator, Kafrelsheikh University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000000230988
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke; Alteplase Adverse Reaction
Keywords: alteplase; hemorragic infarction; Egypt; saudi Arabia; acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: The study consisted of two distinct groups. The first group comprised 464 patients who did not experience hemorrhagic infarction, while the second group comprised 152 patients who experienced hemorrhagic infarction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hemorragic transformation group (Active Comparator): One hundred fifty-two acute ischemic stroke (AIS) patients who had hemorrhagic transformation of brain infarction after 24-36 hours of receiving alteplase.
  Interventions: Drug: Alteplase
- non-hemorragic transformation group (Active Comparator): Four hundred sixty-four acute ischemic stroke (AIS) patients did not have a hemorrhagic transformation of brain infarction after 24-36 hours of receiving alteplase.
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Alteplase — Following the guidelines set by the American Heart Association/American Stroke Association (AHA/ASA), inclusion and exclusion criteria for alteplase were established; 0.9 mg/kg of alteplase up to a maximum dose of 90 mg was administered intravenously to eligible individuals within 4.5 hours of the beginning of their clinical manifestations (10% bolus, 90% infusion in 1 hour). After receiving IV-alteplase, all patients continued their management and rehabilitation in the stroke unit.
  Arms: Hemorragic transformation group
Drug: Alteplase — Following the guidelines set by the American Heart Association/American Stroke Association (AHA/ASA), inclusion and exclusion criteria for alteplase were established; 0.9 mg/kg of alteplase up to a maximum dose of 90 mg was administered intravenously to eligible individuals within 4.5 hours of the beginning of their clinical manifestations (10% bolus, 90% infusion in 1 hour). After receiving IV-alteplase, all patients continued their management and rehabilitation in the stroke unit.
  Arms: non-hemorragic transformation group

SUMMARY:
The investigators evaluated whether the characteristics of ischemic stroke patients, door-to-needle time, and stroke risk factors were predictive variables for different subtypes of post-alteplase hemorrhagic transformation of brain infarction.

DETAILED DESCRIPTION:
Investigators conducted a prospective cohort study between June 2021 and October 2023. They screened 1450 patients who presented with AIS and received alteplase and included 616 AIS patients who met the inclusion criteria and were diagnosed based on a thorough clinical assessment, including a detailed medical history, physical examination, and specific brain imaging results and treated with alteplase within four and half hours of stroke onset.

The investigators assessed the patients' follow-up brain imaging to detect the subtypes of hemorrhagic transformation after receiving alteplase.

The study consisted of two distinct groups. The first group consisted of 464 patients who did not experience hemorrhagic infarction, while the second group comprised 152 patients who experienced hemorrhagic infarction.

The investigators evaluated whether the characteristics of ischemic stroke patients, door-to-needle time, and stroke risk factors were predictive variables for different subtypes of post-alteplase hemorrhagic transformation of brain infarction.

ELIGIBILITY:
Inclusion Criteria:

* The investigators enrolled individuals of both genders, aged between 18 and 75, who presented with acute first-ever ischemic stroke and were eligible for thrombolysis.

Exclusion Criteria:

* The investigators excluded patients who had not been followed up on for 90 days after enrollment,
* Those with alteplase contraindications or did not receive the total dose of alteplase due to any reason were excluded
* The investigators excluded patients with a known history of persistent or recurrent CNS pathology (e.g., epilepsy, meningioma, multiple sclerosis, history of head trauma with a residual neurological deficit).
* The investigators excluded patients who had recurrent ischemic stroke diagnosed by appropriate clinical history and/or MRI brain findings.
* The investigators excluded patients with symptoms of major organ failure, active malignancies, or an acute myocardial infarction within the previous six weeks.
* The investigators also excluded pregnant and lactating patients with stroke due to venous thrombosis and stroke following cardiac arrest

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
predictors of the hemorrhagic infarction type 1 | 48 hours
  The investigators employed univariate and multivariate Logistic regression analysis to assess the ability of patients' characteristics and risk factors to predict hemorrhagic infarction type 1 after 24-36 hours of receiving alteplase after acute ischemic stroke.

SECONDARY OUTCOMES:
predictors of the hemorrhagic infarction type 2 | 48 hours
  The investigators employed univariate and multivariate Logistic regression analysis to assess the ability of patients' characteristics and risk factors to predict hemorrhagic infarction type 1 after 24-36 hours of receiving alteplase after acute ischemic stroke.
predictors of the parenchymal hematoma type 1 | 48 hours
  The investigators employed univariate and multivariate Logistic regression analysis to assess the ability of patients' characteristics and risk factors to predict parenchymal hematoma type 1 after 24-36 hours of receiving alteplase after acute ischemic stroke.
predictors of the parenchymal hematoma type 2 | 48 hours
  The investigators employed univariate and multivariate Logistic regression analysis to assess the ability of patients' characteristics and risk factors to predict parenchymal hematoma type 2 after 24-36 hours of receiving alteplase after acute ischemic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed G. Zeinhom, MD, Principal Investigator — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
All the data supporting this research's findings may be available from the principal investigator, Mohamed G. Zeinhom, upon reasonable request.

REFERENCES:
- [Result] Lopez AD, Mathers CD, Ezzati M, Jamison DT, Murray CJ. Global and regional burden of disease and risk factors, 2001: systematic analysis of population health data. Lancet. 2006 May 27;367(9524):1747-57. doi: 10.1016/S0140-6736(06)68770-9. PMID 16731270
- [Result] Zeinhom MG, Aref HM, El-Khawas H, Roushdy TM, Shokri HM, Elbassiouny A. A pilot study of the ticagrelor role in ischemic stroke secondary prevention. Eur Neurol. 2022;85(1):50-55. doi: 10.1159/000518786. Epub 2021 Aug 30. PMID 34515113
- [Result] Bruno A, Levine SR, Frankel MR, Brott TG, Lin Y, Tilley BC, Lyden PD, Broderick JP, Kwiatkowski TG, Fineberg SE; NINDS rt-PA Stroke Study Group. Admission glucose level and clinical outcomes in the NINDS rt-PA Stroke Trial. Neurology. 2002 Sep 10;59(5):669-74. doi: 10.1212/wnl.59.5.669. PMID 12221155
- [Result] Aref HM, El-Khawas H, Elbassiouny A, Shokri HM, Zeinhom MG, Roushdy TM. A randomized pilot study of the efficacy and safety of loading ticagrelor in acute ischemic stroke. Neurol Sci. 2023 Feb;44(2):765-771. doi: 10.1007/s10072-022-06525-7. Epub 2022 Nov 30. PMID 36446950
- [Derived] Zeinhom MG, Ahmed SR, Kohail AM, Kamel IFM, Abdelrahman AM, Al-Nozha OM, Almoataz M, Youssif TYO, Daabis AMA, Refat HM, Ebied AAMK, Elbassiouny A, Akl AZO, Shuaib A, Ismaiel M, Ibrahem AIDM, Khalil MFE. A multicenter trial on the predictors of different subtypes of hemorrhagic infarction after thrombolysis. Sci Rep. 2024 Nov 30;14(1):29822. doi: 10.1038/s41598-024-76189-0. PMID 39616189